CLINICAL TRIAL: NCT01060046
Title: Analysis and Characterization of in Vivo Tissue Remodeling in Routine Biologic Mesh Explants From Patients Undergoing Reoperation for Recurrent Hernia or Revision of a Prior Surgical Site
Brief Title: Analysis and Characterization of Biologic Implants
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 201101959
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Ventral Hernia; Post-mastectomy Breast Reconstruction
Keywords: biologic mesh; ventral hernia repair; breast reconstruction; MMPs
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy samples of previously implanted biologic meshes, biopsy samples of native abdominal wall fascia
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with previously implanted biologic mesh: All patients undergoing a repeat operation to repair a recurrent hernia or to revise a surgical site which has been previously repaired using a biologic mesh.
- Control patients: Any patient undergoing a surgical procedure where fascial biopsy would not compromise the integrity of the procedure.

SUMMARY:
The purpose of this study is to investigate what happens to biologic mesh in the body over time on a molecular level. To date, it is not known what agents, enzymes, or proteins are interacting at the implantation site that contributes to mesh remodeling and/or degradation. Investigators on this project will identify patients with previously placed mesh who are needing reoperation on the same site and take a biopsy of the mesh during the normal course of surgery. Basic data surrounding the surgical procedure will be collected. The mesh samples will be analyzed for enzymes and proteins and examined histologically for processes that signify remodeling and/or degradation. Control patients will undergo biopsy of abdominal fascia at laparoscopic trocar sites in a manner that will not affect the outcome(s) of their procedure or other risk to the incision site.

DETAILED DESCRIPTION:
Several such biologic meshes have now been developed and marketed for use in hernia repair and soft tissue reconstruction. These biologics include one product derived from porcine intestinal submucosa (SurgisisTM, Cook Medical), another derived from porcine dermis (CollaMendTM, C.R. Bard Inc.) and several others derived from decellularized human dermis, such as AlloDermTM (LifeCell Corp.), AlloMaxTM (C.R. Bard Inc.), and FlexHDTM (Musculoskeletal Transplant Foundation). Although similar in concept and design, each of these biologic meshes is produced in a distinct, proprietary fashion, and different techniques are used by each company in the processing and storage of their respective products. Given that these processing steps are protected industrial intellectual property, rigorous comparison of the performance of each mesh is very difficult. It is expected that certain methods, such as employing or avoiding chemical cross-linking of the ECM proteins, would lead to significant differences in cell migration into, and biochemical remodeling of each individual mesh. These differences may be of particular importance in the scenario of laparoscopic ventral hernia repair, where the mesh is placed in direct apposition to the parietal peritoneum. In this case, if the biologic were to remodel and take on more of the properties of the distensible peritoneum rather than that of the stronger abdominal wall fascia, this could have a significant impact on the long-term strength and durability of the hernia repair. A similar situation could also be foreseen to occur at the esophageal hiatus and/or the site of an intestinal stoma. We feel that it is thus important to study the remodeling processes that these meshes undergo over time and determine if differences in product processing or anatomical position have any effect on mesh incorporation and hernia integrity. Many of these meshes have already been used in human subjects, yet a certain number of these patients are known have suffered hernia recurrences requiring reoperation and removal of some or all of the original mesh prostheses. It is our belief that these biologic explants represent an excellent source of material to study the remodeling process over numerous given time points and at various anatomic locations. We feel it is also important to compare the explanted biologic meshes to "control" tissues, to examine how successfully the biologic meshes are mimicking native tissue at the molecular and histologic level. To eliminate confounding factors, explanted meshes will be compared to biopsies of abdominal wall fascia from patients undergoing non-hernia related surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a repeat operation to repair a recurrent hernia or revise a surgical site which has been previously repaired using one of the aforementioned biologic meshes. Any patient undergoing a surgical procedure where fascial biopsy would not compromise the integrity of the procedure.

Exclusion Criteria:

* For those subjects meeting the inclusion criteria, the only population that will be excluded is that of prisoners.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected from the practices of the surgeons listed on the investigational team.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2007-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent D Matthews, MD, Principal Investigator — Washington University School of Medicine; Corey Deeken, PhD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Buinewicz B, Rosen B. Acellular cadaveric dermis (AlloDerm): a new alternative for abdominal hernia repair. Ann Plast Surg. 2004 Feb;52(2):188-94. doi: 10.1097/01.sap.0000100895.41198.27. PMID 14745271
- [Background] Burger JW, Halm JA, Wijsmuller AR, ten Raa S, Jeekel J. Evaluation of new prosthetic meshes for ventral hernia repair. Surg Endosc. 2006 Aug;20(8):1320-5. doi: 10.1007/s00464-005-0706-4. Epub 2006 Jul 24. PMID 16865616
- [Background] Butler CE, Prieto VG. Reduction of adhesions with composite AlloDerm/polypropylene mesh implants for abdominal wall reconstruction. Plast Reconstr Surg. 2004 Aug;114(2):464-73. doi: 10.1097/01.prs.0000132670.81794.7e. PMID 15277815
- [Background] Butler CE. The role of bioprosthetics in abdominal wall reconstruction. Clin Plast Surg. 2006 Apr;33(2):199-211, v-vi. doi: 10.1016/j.cps.2005.12.009. PMID 16638463
- [Background] Butler CE, Langstein HN, Kronowitz SJ. Pelvic, abdominal, and chest wall reconstruction with AlloDerm in patients at increased risk for mesh-related complications. Plast Reconstr Surg. 2005 Oct;116(5):1263-75; discussion 1276-7. doi: 10.1097/01.prs.0000181692.71901.bd. PMID 16217466
- [Background] Dalla Vecchia L, Engum S, Kogon B, Jensen E, Davis M, Grosfeld J. Evaluation of small intestine submucosa and acellular dermis as diaphragmatic prostheses. J Pediatr Surg. 1999 Jan;34(1):167-71. doi: 10.1016/s0022-3468(99)90250-6. PMID 10022165
- [Background] Diaz S, Brunt LM, Klingensmith ME, Frisella PM, Soper NJ. Laparoscopic paraesophageal hernia repair, a challenging operation: medium-term outcome of 116 patients. J Gastrointest Surg. 2003 Jan;7(1):59-67. doi: 10.1016/S1091-255X(02)00151-8. PMID 12559186
- [Background] Draaisma WA, Gooszen HG, Tournoij E, Broeders IA. Controversies in paraesophageal hernia repair: a review of literature. Surg Endosc. 2005 Oct;19(10):1300-8. doi: 10.1007/s00464-004-2275-3. Epub 2005 Aug 4. PMID 16151684
- [Background] Franklin ME Jr, Gonzalez JJ Jr, Glass JL. Use of porcine small intestinal submucosa as a prosthetic device for laparoscopic repair of hernias in contaminated fields: 2-year follow-up. Hernia. 2004 Aug;8(3):186-9. doi: 10.1007/s10029-004-0208-7. Epub 2004 Feb 26. PMID 14991410
- [Background] Holton LH 3rd, Kim D, Silverman RP, Rodriguez ED, Singh N, Goldberg NH. Human acellular dermal matrix for repair of abdominal wall defects: review of clinical experience and experimental data. J Long Term Eff Med Implants. 2005;15(5):547-58. doi: 10.1615/jlongtermeffmedimplants.v15.i5.70. PMID 16218902
- [Background] Kish KJ, Buinewicz BR, Morris JB. Acellular dermal matrix (AlloDerm): new material in the repair of stoma site hernias. Am Surg. 2005 Dec;71(12):1047-50. PMID 16447477
- [Background] Kolker AR, Brown DJ, Redstone JS, Scarpinato VM, Wallack MK. Multilayer reconstruction of abdominal wall defects with acellular dermal allograft (AlloDerm) and component separation. Ann Plast Surg. 2005 Jul;55(1):36-41; discussion 41-2. doi: 10.1097/01.sap.0000168248.83197.d4. PMID 15985789
- [Background] Miller RS, Morris JA Jr, Diaz JJ Jr, Herring MB, May AK. Complications after 344 damage-control open celiotomies. J Trauma. 2005 Dec;59(6):1365-71; discussion 1371-4. doi: 10.1097/01.ta.0000196004.49422.af. PMID 16394910
- [Background] Oelschlager BK, Barreca M, Chang L, Pellegrini CA. The use of small intestine submucosa in the repair of paraesophageal hernias: initial observations of a new technique. Am J Surg. 2003 Jul;186(1):4-8. doi: 10.1016/s0002-9610(03)00114-4. PMID 12842738
- [Background] Oelschlager BK, Pellegrini CA, Hunter J, Soper N, Brunt M, Sheppard B, Jobe B, Polissar N, Mitsumori L, Nelson J, Swanstrom L. Biologic prosthesis reduces recurrence after laparoscopic paraesophageal hernia repair: a multicenter, prospective, randomized trial. Ann Surg. 2006 Oct;244(4):481-90. doi: 10.1097/01.sla.0000237759.42831.03. PMID 16998356
- [Background] Scott BG, Welsh FJ, Pham HQ, Carrick MM, Liscum KR, Granchi TS, Wall MJ Jr, Mattox KL, Hirshberg A. Early aggressive closure of the open abdomen. J Trauma. 2006 Jan;60(1):17-22. doi: 10.1097/01.ta.0000200861.96568.bb. PMID 16456431
- [Background] Silverman RP, Li EN, Holton LH 3rd, Sawan KT, Goldberg NH. Ventral hernia repair using allogenic acellular dermal matrix in a swine model. Hernia. 2004 Dec;8(4):336-42. doi: 10.1007/s10029-004-0241-6. PMID 15185131
- [Derived] Cavallo JA, Roma AA, Jasielec MS, Ousley J, Creamer J, Pichert MD, Baalman S, Frisella MM, Matthews BD, Deeken CR. Remodeling characteristics and collagen distribution in biological scaffold materials explanted from human subjects after abdominal soft tissue reconstruction: an analysis of scaffold remodeling characteristics by patient risk factors and surgical site classifications. Ann Surg. 2015 Feb;261(2):405-15. doi: 10.1097/SLA.0000000000000471. PMID 24374547